CLINICAL TRIAL: NCT01206920
Title: Development of a City-Wide Cohort of HIV-Infected Persons in Care in the District of Columbia: The DC Cohort
Brief Title: The DC Cohort Longitudinal HIV Status Neutral Study
Acronym: DC Cohort
Status: Recruiting | Type: Observational
Sponsor: George Washington University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Amanda D. Castel, PI, George Washington University
Other Study IDs: 071029; R24AI152598 (NIH)
Record Dates: First submitted 2010-09-21; First posted 2010-09-22 (Estimated); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: HIV; AIDS
Keywords: HIV; AIDS; Co-morbidities
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Treatment Cohort: These are individuals who are diagnosed with HIV and receiving care at a participating DC Cohort clinical site.
- Prevention Cohort: These are individuals who are receiving HIV preventive services at a participating DC Cohort site.

SUMMARY:
The goal of the DC Cohort is to establish a clinic-based city-wide longitudinal cohort that will describe clinical outcomes, and improve the quality of care for patients diagnosed with Human Immunodeficiency Virus/Acquired Immune Deficiency Syndrome (HIV/AIDS) or at higher risk for acquiring HIV and receiving care in Washington, DC.

DETAILED DESCRIPTION:
All major community and academic clinics treating persons with HIV in the District of Columbia (DC) are included in the "DC Cohort", with consideration to be given subsequently to the inclusion of large private physician practices. Recruitment of persons at higher risk for acquiring HIV will occur in selected clinics based on the numbers of persons estimated to be receiving HIV preventive services at those clinics. Socio-demographics, risk factors, treatments, diagnoses, labs and procedures documented in outpatient medical record systems will be included in the DC Cohort database. Routine reports will be generated every quarter for sites comparing their participants' socio-demographics, clinical status, treatments, and outcomes to all other data in the DC Cohort database, and other comparisons specifically requested by sites. All sites will be provided analytic support in research areas of interest.

ELIGIBILITY:
Treatment Cohort Inclusion Criteria:

* Patient is receiving care for HIV at one or more of the twelve participating clinics in the DC Cohort.
* Patient is either age 18 years or older, or seeks HIV care independently and is able to understand and sign informed consent.
* Patient is a minor who is consented by a parent or legal guardian.

Treatment Cohort Exclusion Criteria:

* Patient is unable or refuses to provide informed consent.
* Minor children ages 12 through 17 who are unaware of their HIV status

Prevention Cohort Inclusion Criteria:

Persons receiving any antiretroviral prescription without evidence of HIV or Hepatitis B infection

* PrEP (e.g., TDF/FTC, Descovy, Apretude)
* Combination ART indicative of nPEP in an HIV-uninfected person
* Persons receiving an antiretroviral prescription indicative of DoxyPEP Doxycycline 200mg PO taken within 72 hrs of unprotected sexual encounter (or variations thereof where clearly not prescribed as a treatment course)
* Test positive for ≥1 bacterial STI (positive gonorrhea (GC/NG) or chlamydia (CT) test or positive syphilis test requiring treatment within one year)

  * 2 bacterial STI (GC, chlamydia, syphilis) tests at 2 or more different encounters
  * 2 HIV tests at 2 or more different encounters
* Patient requesting PrEP at their clinical visit
* Patient requesting nPEP at their clinical visit
* People who identify as injecting drugs

Patients with a Z29.81 Encounter for HIV pre-exposure prophylaxis

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Study participants will include men, women and children receiving HIV prevention, care or treatment services at major publicly-funded, government and academic medical centers in the District of Columbia.
Sampling Method: Non-Probability Sample
Enrollment: 19000 (Estimated)
Dates: Start 2011-01 (Actual); Primary Completion 2041-01 (Estimated); Study Completion 2041-01 (Estimated)

PRIMARY OUTCOMES:
viral suppression among persons with HIV | through study completion, an average of 10 years from enrollment to the end of study follow up
  The study will assess rates of viral suppression (defined as an HIV RNA test less than 200 copies/ml) from enrollment to 10 years post enrollment.
clinical outcomes persons at higher risk for acquiring HIV | through study completion, an average of 5 years from enrollment to the end of study follow up period
  Persons who are receiving HIV preventive services will be followed longitudinally to assess time to HIV positivity from baseline to 5 years post enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Amanda D Castel, MD, MPH, Principal Investigator — George Washington University
Locations (14):
- United States (14):
  - Kaiser Permanente Mid-Atlantic States, Washington D.C., District of Columbia
  - Unity Health Care, Washington D.C., District of Columbia
  - Georgetown University, Washington D.C., District of Columbia
  - La Clinica Del Pueblo, Washington D.C., District of Columbia
  - Whitman-Walker Health, Washington D.C., District of Columbia
  - Children's National Medical Center--Pediatric Clinic, Washington D.C., District of Columbia
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Washington Health Institute, Washington D.C., District of Columbia
  - Family and Medical Counseling Service, Washington D.C., District of Columbia
  - George Washington Medical Faculty Associates, Washington D.C., District of Columbia
  - Howard University Hospital--Adult Clinic, Washington D.C., District of Columbia
  - Howard University Hospital--Pediatric Clinic, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center, Washington D.C., District of Columbia
  - Us Helping Us, People into Living, Inc., Washington D.C., District of Columbia

REFERENCES:
- See also: DC Cohort Website — http://go.gwu.edu/dccohort